CLINICAL TRIAL: NCT05717465
Title: Communicating Risks: Consent for Lumbar Puncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Anand S. Pandit, Neurosurgical Specialty Registrar (ST4), University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 21837.001
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Informed Consent, Health Literacy, Risk, Spinal Puncture, Neurosurgery
Keywords: Health Literacy; Risk; Spinal Puncture

STUDY DESIGN:
Intervention Model Description: Upon clicking the link to the study questionnaire, participants were randomized to either receive the control or intervention questionnaire. This was done through Qualtrics (Qualtrics, Provo, UT) built-in randomization.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators were blind as to which arm participants were allocated to as the randomization and intervention/control exposure occurs after participants open the link to the study questionnaire. The same link would allocate participants to either the control/intervention group.
  Outcomes were assessed within the questionnaire without any human input No care providers were present in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard informed consent (Active Comparator): Video with audio narration containing information provided in the standard informed consent process for a lumbar puncture
  Interventions: Other: Standard informed consent
- Visual aid group (Experimental): Video with identical audio narration (to the control) containing information provided in the standard informed consent process for a lumbar puncture. The video also received statistical information in the form of visual aids; anatomy diagrams, Paling diagrams and Paling scales
  Interventions: Other: Anatomy diagrams; Other: Standard informed consent

INTERVENTIONS:
Other: Anatomy diagrams — The visual aids used included:
  * An anatomical diagram illustrating how a lumbar puncture is carried out
  * Paling palette, diagram illustrating the number of individuals affected by a particular condition
  * Paling perspective scale, diagram comparing the risk of an event occurring in comparison to other 'everyday' risks
  Other Names: Paling diagrams; Paling scale
  Arms: Visual aid group
Other: Standard informed consent — Audio narration of a video containing text information relating to the lumbar puncture procedure (including risks) and an image of a consent form

SUMMARY:
The goal of this randomized control trial is to compare the effect of visual aids on the recall of probabilistic risks in healthy participants. The main questions it aims to answer are:

* Will participants consented using a consent process incorporating visual aids recall the consent process better?
* Will participants consented with a consent process incorporating visual aids have higher acceptability if a hypothetical, simulated complication were to occur?
* Is this method of consent (visual aids) usable, appropriate and acceptable? Participants will be required to watch a brief video containing information on how a lumbar puncture is performed as well as the associated risks.
* Participants in the intervention group will receive information in the form of various visual aids (e.g. anatomical diagrams, paling palettes and paling perspective scales). The audio narration and information provided in both groups is identical.
* Participants will be tested on their knowledge of the procedure
* Participants will be asked to rate their response to a series of procedure specific statements and statements from other validated scales.

Researchers will compare the control and intervention group to see if there is improvement in the recall of information and which consent process is more acceptable, appropriate and usable.

DETAILED DESCRIPTION:
Background:

Informed consent is an essential process in clinical decision-making, through which healthcare providers educate patients about the benefits, risks and alternatives of a given procedure or intervention in a descriptive way. An accurate understanding of the numerical information pertaining to risk is important because individuals perceive probability differently while also having different thresholds for what they would consider an unacceptable. This is vital for shared decision making to ensure that patients only undergo procedures or treatments where their understanding of the risks is in line with their personal level of acceptability. Aid tools have been employed to elaborate and communicate probabilistic risk information in areas such as screening (1). To the best of our knowledge there are no studies which evaluate the application of such visual aids on probabilistic information in surgical patients.

Objectives:

Our study aims to explore the effectiveness of visual aids to help communicate statistical information during the informed consent of a common clinical procedure: a lumbar puncture. We compare the effectiveness of this enhanced consent process against a typical consent method without visual aids

Methods:

Healthy participants were recruited within our institution and randomized using Qualtrics to complete a questionnaire containing either the control video or intervention video. Both videos contained identical audio narration however the intervention video included additional visual aids.

Status:

Recruitment of participants has been completed and the study has been written-up and submitted for publication and presentations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Above 18 years old
* No underlying cognitive impairment

Exclusion Criteria:

* Individuals with prior experience receiving, performing or observing a lumbar puncture
* Lacks capacity
* Hospitalized individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-03-27 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Recall of probabilistic risk | Measured immediately following exposure to control/intervention
  Measured by the number of correct answers to our procedure specific questionnaire

SECONDARY OUTCOMES:
Response to procedure specific statements | Measured immediately following exposure to control/intervention
  Measured using 5-point likert scale responses
Acceptability | Measured immediately following exposure to control/intervention
  Measured by the Acceptability of Intervention Measure (AIM) scale
Approrpiateness | Measured immediately following exposure to control/intervention
  Measured by the Intervention Appropriateness Measure (IAM) scale
Usability | Measured immediately following exposure to control/intervention
  Measured by the System Usability Scale (SUS)

CONTACTS AND LOCATIONS:
Overall Officials: Anand S Pandit, PhD MRCS, Principal Investigator — University College London/University College London Hospital; Hani J Marcus, PhD FRCS (SN), Principal Investigator — University College London/University College London Hospital
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coyle M, Gillies K. A systematic review of risk communication in clinical trials: How does it influence decisions to participate and what are the best methods to improve understanding in a trial context? PLoS One. 2020 Nov 16;15(11):e0242239. doi: 10.1371/journal.pone.0242239. eCollection 2020. PMID 33196663